CLINICAL TRIAL: NCT05147753
Title: Effects of Moxonidine Administration on Serum Neuropeptide Y Levels in Hypertensive Individuals: A Prospective Observational Study
Brief Title: Moxonidine Effects on Neuropeptide Y
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Prof. Triantafyllos Didangelos, Associate Professor of Internal Medicine-Diabetology, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7337_20042021
Record Dates: First submitted 2021-11-18; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Hypertension
Keywords: hypertension; obesity; Neuropeptide Y; moxonidine
MeSH Terms: conditions — Obesity; Hypertension | interventions — moxonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Experimental): 0.6 mg moxonidine daily
  Interventions: Drug: Moxonidine

INTERVENTIONS:
Drug: Moxonidine — 0.6 mg moxonidine daily

SUMMARY:
Treatment with monotherapy of moxonidine 0.6 mg daily in treatment-naïve subjects with mild or moderate hypertension

DETAILED DESCRIPTION:
Treatment with 0.6 mg moxonidine daily in treatment-naïve subjects with mild or moderate hypertension according to guidelines (Stage 1: Systolic Blood Pressure =140-159 mmHg, Diastolic Blood Pressure =90-99 mmHg, and Stage 2: systolic blood pressure=160-179 mmHg, diastolic blood pressure=100-109 mmHg) that require monotherapy and reevaluation after 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* treatment-naïve subjects with mild or moderate hypertension according to Joint National Committee 7 and European Society Hypertension / European Society Cardiology 2008 (Stage 1: Systolic Blood Pressure =140-159 mmHg, Diastolic Blood Pressure =90-99 mmHg, and Stage 2: Systolic=160-179 mmHg, Diastolic=100-109 mmHg) that require monotherapy

Exclusion Criteria:

* age beyond 25-75 years,
* not taking currently anti-hypertensive medication
* not taking anti-diabetic or lipid lowering medication and other diseases or conditions that may influence blood pressure, heart rate and catecholamines' and Neuropeptide Y levels, including anemia, fever, stage III hypertension, coronary artery disease, recent (less than 6 months) myocardial infraction or stroke, heart failure, secondary hypertension, diabetes mellitus, abnormal thyroid status or other obesity-related endocrinopathies, pregnancy, kidney failure, alcohol abuse, malignancies, depression or other psychiatric illnesses, such as schizophrenia,

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01-11 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
serum Neuropeptide Y levels | 12 weeks
  ELISA
systolic blood pressure | 12 weeks
  mmHg
diastolic blood pressure | 12 weeks
  mmHg

SECONDARY OUTCOMES:
Weight | 12 weeks
  kg
Body Mass Index | 12 weeks
  kg/m2
Total Cholesterol | 12 weeks
  mg/dl
HDL Cholesterol | 12 weeks
  mg/dl
LDL Cholesterol | 12 weeks
  mg/dl
Serum triglycerides | 12 weeks
  mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Karlafti, MD, PhD, Principal Investigator — AHEPA University Hospital

IPD SHARING:
Plan to Share IPD: No